CLINICAL TRIAL: NCT06281158
Title: A Study of the Pharmacokinetics of [14C]-DNL343 Following a Single Oral Dose in Healthy Male Participants
Brief Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-DNL343 Following a Single Oral Dose in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-F-0009
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C-DNL343 (Experimental)
  Interventions: Drug: [14C]-DNL343

INTERVENTIONS:
Drug: [14C]-DNL343 — Single dose

SUMMARY:
This is a Phase 1, open-label, nonrandomized, single-dose study in healthy male participants to investigate the absorption, metabolism and excretion of DNL343.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged between 18 to 65 years, inclusive
* Body mass index between 18.0 and 32.0 kg/m2
* In good health
* When engaging in sex with a woman of child bearing potential, both the male participant and his female partner must use highly effective contraception
* History of a minimum of 1 bowel movement per day

Exclusion Criteria:

* History or clinical manifestation of any clinically significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Have a history of malignancy, except fully resected basal cell carcinoma
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Have previously completed or withdrawn from this study or any other study investigating DNL343 and have previously received DNL343

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
PK Parameter: AUC0-∞ | 28 days
  The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL343 in plasma
PK Parameter: AUC0-tlast | 28 days
  Area under the concentration-time curve from time zero to the last quantifiable time point (AUC0-tlast) of DNL343 in plasma
PK Parameter: Cmax | 28 days
  Maximum observed concentration (Cmax) of DNL343 in plasma
PK Parameter: Tmax | 28 days
  Time to maximum observed concentration (Tmax) of DNL343 in plasma
PK Parameter: t1/2 | 28 days
  Terminal elimination half-life (t1/2) of DNL343 in plasma
Total radioactivity in plasma and whole blood | 28 days
Total radioactivity in blood-to-plasma ratio | 28 days
Extent and rate of recovery of total radioactivity in urine and feces | 28 days

SECONDARY OUTCOMES:
PK Parameter: AUC0-∞ | 28 days
  The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of a DNL343 metabolite in plasma
PK Parameter: AUC0-tlast | 28 days
  Area under the concentration-time curve from time zero to the last quantifiable time point (AUC0-tlast) of a DNL343 metabolite in plasma
PK Parameter: Cmax | 28 days
  Maximum observed concentration (Cmax) of a DNL343 metabolite in plasma
PK Parameter: Tmax | 28 days
  Time to maximum observed concentration (Tmax) of a DNL343 metabolite in plasma
PK Parameter: t1/2 | 28 days
  Terminal elimination half-life (t1/2) of a DNL343 metabolite in plasma
DNL343 and a DNL343 metabolite recoveries in urine | 28 days
Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Claire Meyer, MD, Study Director — Denali Therapeutics
Locations (1):
- Clinical Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No